CLINICAL TRIAL: NCT05027724
Title: Technology Assisted Solutions for the Recognition of Objective Physiological Indicators of Post-Coronavirus-19 Fatigue
Acronym: TROPIC
Status: Completed | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Science Foundation Ireland (Other)
Responsible Party: Principal Investigator, Román Romero Ortuño, Associate Professor, Discipline of Medical Gerontology, Trinity College Dublin, University of Dublin, Trinity College
Other Study IDs: 20/COV/8493
Record Dates: First submitted 2021-08-23; First posted 2021-08-30 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Covid19; Post Viral Fatigue
Keywords: fatigue; deconditioning; orthostatic intolerance; long-COVID
MeSH Terms: conditions — COVID-19; Fatigue; Orthostatic Intolerance; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preliminary research from our group indicates that up to half of COVID-19 patients are experiencing symptoms consistent with severe fatigue a median of 10 weeks after their initial illness, while almost one third of those previously employed have not returned to work. At present, most clinical and research measurements of fatigue have relied upon self-reported perception of sensations such as exhaustion or weariness. Using such tools, there is an inherent challenge for clinicians in differentiating between patients who are experiencing fatigue at a psychosocial level, versus those who are actively physiologically and neurocognitively deconditioned. The TROPIC study will use our existing clinical expertise and technology assisted solutions to address features of post-COVID-19 fatigue by quantifying physiological signatures of adverse sequelae in adult patients previously diagnosed with COVID-19, who are now COVID-19 negative. Our suite of assessments will encompass four systems; physical deconditioning, orthostatic instability, neurocognitive deficits and respiratory sequelae. This will not only inform accurate objective diagnostics of post-COVID-19 Chronic Fatigue Syndrome, but will also guide clinicians in directing the most appropriate therapeutic interventions with maximum efficacy and specificity, bringing not only patient-related but also health system and economic benefits.

DETAILED DESCRIPTION:
Background: At the time of writing, over 214 million people globally are infected with the Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). It is estimated that up to 50% of people are experiencing debilitating levels of fatigue months after recovering from the acute phase of COVID-19, known as post COVID-19 Chronic Fatigue Syndrome (CFS). The most challenging aspect in the management of CFS for clinicians is the lack of objective measurement tools. At present, most clinical and research measurements of fatigue have relied upon self-reported perceptions of sensations such as exhaustion or weariness. We believe that an objective, technology-based assessment of this complex condition is required for the quantification of complex multi-system dynamic physiological signals in order to guide clinicians in directing targeted valuable resources towards therapeutic interventions with specificity and rigour to those patients who are most in need.

Aim: The aim of the TROPIC study is to identify bio- signals and contributing factors in the development of post-Covid-19 Chronic Fatigue Syndrome using a suite of technology-assisted assessment techniques.

TROPIC STUDY PARTICULARS:

The primary endpoint will be successful recruitment and completion of data collection of 100 participants in the TROPIC cohort.

Setting: Assessments will take place in the Falls and Syncope Unit and Clinical Research Facility of St James's Hospital.

Participants: Participants will be recruited from five sources; (i) the Robert Mayne Day Hospital, (ii) the Falls and Syncope Unit, (iii) Advocacy Groups, (iv) staff who contracted COVID-19, and (v) the Post COVID-19 outpatient (OPD) Clinic.

Participants must be aged 18 years or older, have a history of COVID-19 and be free of exclusion criteria outlined in later sections.

Data collection and analysis: Participants will be invited for one assessment session to St James's Hospital (SJH), where they will undergo a series of neurocardiovascular, neurocognitive and physical performance tests, outlined in more detail in later sections.

ELIGIBILITY:
Inclusion Criteria:

1. Participants age 18 years or over.
2. Able to give informed consent
3. Good spoken and written English
4. History of COVID-19 and experiencing prolonged symptoms.
5. Community ambulant
6. Able to mobilise independently (with or without aid).
7. Able to transfer with minimal assistance of one person from lying to standing.
8. Patients with a history of COVID-19 who now present with a negative swab

Exclusion Criteria:

1. Unwilling to participate
2. Aged less than 18
3. Persons with cognitive impairment / dementia that would render them unable to give informed consent.
4. Persons who are pregnant
5. Persons who require more than min assistance of one person to transfer from lying to standing.
6. Persons who are not independently mobile.
7. Persons with an acute illness.
8. Participants with skin allergies to adhesive tapes.
9. Participants with upper limb lymphoedema (cuff-site)
10. Participants registered as blind or partially blind.
11. Persons for whom tilt testing and exercise testing is contra-indicated as per results of the Physical Activity Readiness Questionnaire or anyone falling under the absolute contra-indications to exercise testing as per the American Heart Association's Guidelines for Exercise testing, including: 1. Acute myocardial infarction within 2 days (or any other acute cardiac event) 2. Unstable angina 3. Uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise 4. Uncontrolled symptomatic heart failure 5. Symptomatic sever aortic stenosis 6. Suspected or known dissecting aneurysm 7. Acute myocarditis or pericarditis 8. Acute pulmonary embolus or pulmonary infarction 9. Acute systemic infection, accompanied by fever, body aches or swollen lymph glands, 10. patients in whom low organ perfusion pressures may compromise end artery supplied tissue, 11 severe left ventricular outflow obstruction, 12. critical mitral stenosis.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants over 18 years, with a history of COVID-19 who are community ambulant, mobilizing independently and free from contra-indications to testing procedures.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Active Stand with Near Infrared Spectroscopy and Electromyography | Day 0
  10 minute supine rest, followed by a three minute stand
Drug Free Passive Head Up Tilt Test | Day 0
  10 minute supine rest, followed by a 10 minute 70 degree passive tilt.
Cardiorespiratory fitness test | Day 0
  Submaximal (Test terminated at 85% maximal heart rate) cycle ergometer based assessment, using indirect calorimetry and heart rate monitoring to determine breath-by-breath oxygen consumption
Gait assessment via Gaitrite™ system | Day 0
  Three walks on a sensor-embedded 9m floor mat. Walk 1 - normal gait Walk 2 - normal gait with dual cognitive task Walk 3 - fast walk
Neurocognitive assessments | Day 0
  Deary-Liewald Task
Strength assessments: leg press and dynamometry | Day 0
  5 times sit-to-stand hand dynamometry based grip strength assessment

SECONDARY OUTCOMES:
Fatigue | Day 0
  Chalder Fatigue Scale (11-item scale with a 0-3 Likert scale for each item. Scores range from 0 - 33. A higher score represents more severe fatigue)
Depression | Day 0
  Center for Epidemiological Studies-Depression Scale (20-item measure with a 0-3 Likert scale response for each item. Scores range from 0-60. A higher score represents more severe depressive symptoms)
Post-Traumatic Stress (after contracting COVID-19) | Day 0
  Impact of Events Scale (Revised) (22-item questionnaire with a 0-5 Likert scale for each response. Scores range from 0 - 110. A higher score indicates an increased perception of stress after an event).

CONTACTS AND LOCATIONS:
Overall Officials: Roman Romero-Orthuno, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- St James's Hospital, Dublin, Co. Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romero-Ortuno R, Jennings G, Xue F, Duggan E, Gormley J, Monaghan A. Predictors of Submaximal Exercise Test Attainment in Adults Reporting Long COVID Symptoms. J Clin Med. 2022 Apr 23;11(9):2376. doi: 10.3390/jcm11092376. PMID 35566502
- [Derived] Monaghan A, Jennings G, Xue F, Byrne L, Duggan E, Romero-Ortuno R. Orthostatic Intolerance in Adults Reporting Long COVID Symptoms Was Not Associated With Postural Orthostatic Tachycardia Syndrome. Front Physiol. 2022 Mar 4;13:833650. doi: 10.3389/fphys.2022.833650. eCollection 2022. PMID 35309052